CLINICAL TRIAL: NCT01946191
Title: Maintaining Activity and Nutrition Through Technology-Assisted Innovation in Primary Care
Brief Title: Computer-Based Weight Maintenance in Primary Care
Acronym: MAINTAIN-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathleen McTigue, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R18HS021162 (AHRQ)
Record Dates: First submitted 2013-09-16; First posted 2013-09-19 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Body Weight; Weight Loss; Motor Activity
Keywords: Weight maintenance; Electronic health record; Primary care
MeSH Terms: conditions — Body Weight; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coaching Group (Experimental): * 24 months of personalized coaching through the EHR patient portal, with 24 scheduled contacts
  * Online self-monitoring
  * Real-time updates to primary care physicians
  Interventions: Behavioral: 24 months of personalized coaching through the EHR patient portal, with 24 scheduled contacts.; Behavioral: Online self-monitoring; Behavioral: Real-time updates to Primary Care physicians
- Tracking Group (Active Comparator): -Online self-monitoring
  Interventions: Behavioral: Online self-monitoring

INTERVENTIONS:
Behavioral: 24 months of personalized coaching through the EHR patient portal, with 24 scheduled contacts. — Participants were assigned to a specific coach, who contacted the participants via the EHR weekly for 1 month, biweekly in months 2 to 6, monthly in months 7 to 12, and quarterly in months 13 to 24, for a total of 24 scheduled contacts. Coaching group participants received brief questionnaires relevant to weight management, including a text field where they could discuss questions or barriers. On the basis of participant responses and self-monitoring data in the EHR flow sheets, coaches wrote a brief personalized note with advice on questionnaire topics and responses to any queries or barriers mentioned by the participant. Coaching participants who did not complete questionnaires or log information into the flow sheet for 2 weeks were considered inactive and were contacted by telephone or e-mail and invited to reengage at any time. Coaching participants were able to send secure messages to the coach.
  Arms: Coaching Group
Behavioral: Online self-monitoring — Participants were encouraged to log in daily and enter data on weight, diet, and physical activity.
Behavioral: Real-time updates to Primary Care physicians — Referring PCPs of coaching group participants received regular support, including real-time progress reports with counseling tips delivered via the EHR, notification of weight change in increments of at least 10 pounds, and annual progress reports at 12 and 24 months.
  Arms: Coaching Group

SUMMARY:
This randomized trial tested the hypothesis that there would be an incremental benefit of personalized coaching and PCP support in an EHR-based intervention designed to help primary care patients maintain recent intentional weight loss of at least 5%.

DETAILED DESCRIPTION:
MAINTAIN-pc (Maintaining Activity and Nutrition through Technology-Assisted Innovation in Primary Care) was a randomized trial conducted in coordination with practices affiliated with the University of Pittsburgh Medical Center (UPMC). Participants were recruited between October 2013 and February 2015, and follow-up was completed in March 2017. The University of Pittsburgh Institutional Review Board approved the study, and all participants provided written informed consent.

Participants were randomly assigned to EHR tools (tracking group) versus EHR tools plus coaching (coaching group). The EHR tools included weight, diet, and physical activity tracking flow sheets; standardized surveys; and reminders. Participants in the coaching group received 2 years of personalized health coaching through the EHR patient portal. Three study coaches had backgrounds in nursing, nutrition, and exercise physiology. The other 2 received EHR training, and all received training on the study protocol. Participants were assigned to a specific coach, who contacted the participants via the EHR weekly for 1 month, biweekly in months 2 to 6, monthly in months 7 to 12, and quarterly in months 13 to 24, for a total of 24 scheduled contacts. Coaching group participants received brief questionnaires relevant to weight management, including a text field where they could discuss questions or barriers. On the basis of participant responses and self-monitoring data in the EHR flow sheets, coaches wrote a brief personalized note with advice on questionnaire topics and responses to any queries or barriers mentioned by the participant. Coaching participants who did not complete questionnaires or log information into the flow sheet for 2 weeks were considered inactive and were contacted by telephone or e-mail and invited to reengage at any time. Coaching participants were able to send secure messages to the coach. Tracking group participants received questionnaires related to general health promotion (for example, vaccines) each quarter but received no feedback on questionnaire responses or flow sheet entries.

Referring PCPs of coaching group participants received regular support, including real-time progress reports with counseling tips delivered via the EHR, notification of weight change in increments of at least 10 pounds, and annual progress reports at 12 and 24 months. The progress reports were developed using feedback from PCPs and consisted of a 1-page summary of participant weight (current, trajectory, and goal), status in the program (active or inactive), use of study flow sheets (with data if available), and brief subjective comments from the coach. Reports were delivered to the PCP via the EHR within 48 hours before scheduled office visits. An electronic copy was also sent to the participant. Referring PCPs of tracking group participants received annual progress reports at 12 and 24 months. Information about the development of the intervention and the coaching protocol has been published previously

The trial was initially designed to be a 36-month intervention, with the primary outcome defined as weight change at 36 months. Delays in EHR build and recruitment resulted in a decision after enrollment was completed to shorten the intervention to 24 months, with 24-month weight change as the revised primary outcome. In addition, we added an exploratory 30-month weight outcome to assess the duration of effect after the intervention ended. An updated institutional review board protocol (with revised consent) was approved on 25 September 2015. These changes were made before any data were analyzed.

In the result section, we are reporting all pre-specified outcomes unintentionally omitted in the original ClinicalTrials submission.

ELIGIBILITY:
Eligibility criteria included age 18 to 75 years, body mass index (BMI) of 25 kg/m2 or higher, intentional weight loss of at least 5% in the previous 2 years, access to an Internet-connected computer, and receipt of outpatient care from a UPMC PCP.

Exclusion criteria included a medical explanation for recent weight loss (for example, cancer), active preparation for bariatric surgery, bariatric surgery in the previous 5 years, or pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M McTigue, MD, MPH, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- Center for Research on Health Care, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested by researchers after the completion of the primary endpoint publication by contacting Dr. Conroy.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Conroy MB, Bryce CL, McTigue KM, Tudorascu D, Gibbs BB, Comer D, Hess R, Huber K, Simkin-Silverman LR, Fischer GS. Promoting weight maintenance with electronic health record tools in a primary care setting: Baseline results from the MAINTAIN-pc trial. Contemp Clin Trials. 2017 Mar;54:60-67. doi: 10.1016/j.cct.2017.01.001. Epub 2017 Jan 12. PMID 28089764
- [Result] Gibbs BB, Tudorascu D, Bryce CL, Comer D, Fischer GS, Hess R, Huber KA, McTigue KM, Simkin-Silverman LR, Conroy MB. Diet and Physical Activity Behaviors in Primary Care Patients with Recent Intentional Weight Loss. Transl J Am Coll Sports Med. 2017;2(18):114-121. Epub 2017 Sep 15. PMID 29130068
- [Result] Conroy MB, McTigue KM, Bryce CL, Tudorascu D, Gibbs BB, Arnold J, Comer D, Hess R, Huber K, Simkin-Silverman LR, Fischer GS. Effect of Electronic Health Record-Based Coaching on Weight Maintenance: A Randomized Trial. Ann Intern Med. 2019 Dec 3;171(11):777-784. doi: 10.7326/M18-3337. Epub 2019 Nov 12. PMID 31711168
- [Derived] Gibbs BB, Tudorascu D, Bryce CL, Comer D, Fischer GS, Hess R, Huber KA, McTigue KM, Simkin-Silverman LR, Conroy MB. Lifestyle Habits Associated with Weight Regain After Intentional Loss in Primary Care Patients Participating in a Randomized Trial. J Gen Intern Med. 2020 Nov;35(11):3227-3233. doi: 10.1007/s11606-020-06056-x. Epub 2020 Aug 17. PMID 32808209

RESULTS

PARTICIPANT FLOW:
Groups:
- Continued Group: * 24 months of personalized coaching through the EHR patient portal, with 24 scheduled contacts
  * Online self-monitoring
  * Real-time updates to primary care physicians
- Tracking Group: Online self-monitoring
Period: Allocation
Arm/Group | Continued Group | Tracking Group
Started | 98 | 96
Completed | 97 | 95
Not Completed | 1 | 1
Not completed — Did not complete orientation | 1 | 1
Period: Follow-Up, 24-mo Endpoint
Arm/Group | Continued Group | Tracking Group
Started | 97 | 95
Completed | 80 | 77
Not Completed | 17 | 18
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 13 | 15
Period: Primary Outcome Analysis
Arm/Group | Continued Group | Tracking Group
Started | 98 | 95
Completed | 80 (Weight data at 24 months) | 77 (Weight data at 24 months)
Not Completed | 18 | 18

BASELINE CHARACTERISTICS:
Groups:
- Coaching Group: Online self-monitoring along with health coach electronic communication and support and real-time updates to primary care physicians
  Health coach electronic communication and support: Health coach reviews responses to weight-related surveys and provides feedback and advice
  Online self-monitoring: Tracking weight, calories, fat grams, and physical activity in electronic personal health record
  Real-time updates to Primary Care physicians: Primary care physicians will receive updates through electronic health record system before each scheduled appointment
- Tracking Group: Online self-monitoring
  Online self-monitoring: Tracking weight, calories, fat grams, and physical activity in electronic personal health record
- Total: Total of all reporting groups
Arm/Group | Coaching Group | Tracking Group | Total
Number analyzed (Participants) | 98 | 96 | 194
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 84 | 75 | 159
  >=65 years | 14 | 21 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (12) | 53.5 (12.4) | 53.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 76 | 143
  Male | 31 | 20 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 88 | 83 | 171
  Unknown or Not Reported | 9 | 11 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 11 | 19
  White | 88 | 83 | 171
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 98 | 96 | 194
Non-smoker [Count of Participants; unit: Participants] | 95 | 94 | 189
Education post high school [Count of Participants; unit: Participants] | 95 | 90 | 185
Weight [Mean (Standard Deviation); unit: kg] | 88.2 (18.7) | 83.3 (19.2) | 85.8 (19.1)
Waist circumference [Mean (Standard Deviation); unit: cm] | 99.7 (13.9) | 96.2 (16.8) | 97.9 (15.5)
Any moderate physical activity [Count of Participants; unit: Participants] — Moderate and vigorous physical activity are the n (%) of participants reporting any of each type of PA on the baseline BRFSS physical activity survey
  Participants | 93 | 92 | 185
Any vigorous physical activity [Count of Participants; unit: Participants] — Moderate and vigorous physical activity are the n (%) of participants reporting any of each type of PA on the baseline BRFSS physical activity survey
  Participants | 59 | 60 | 119
High cholesterol [Count of Participants; unit: Participants] | 46 | 37 | 83
Hypertension [Count of Participants; unit: Participants] | 56 | 40 | 96
Arthritis (Knee and/or Hip) [Count of Participants; unit: Participants] | 30 | 28 | 58
Diabetes or Pre-Diabetes [Count of Participants; unit: Participants] | 20 | 22 | 42
Anxiety/Depression [Count of Participants; unit: Participants] | 30 | 23 | 53
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 124.7 (14.2) | 121.6 (13.0) | 123.2 (13.7)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 75.4 (8.9) | 72.7 (10.1) | 74.0 (9.6)

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: Weight (kg), change from baseline, Estimate (SE) [95% confidence interval]
Time Frame: Baseline to 24 months
Measure: Mean (Standard Error); unit: kg
Arm/Group | Coaching Group | Tracking Group
Number analyzed (Participants) | 80 | 77
kg | 2.07 (0.62) | 4.93 (0.63)

2. Secondary Outcome: BMI
Description: Body Mass Index, change from baseline, Estimate (SE) [95% CI]
Time Frame: Baseline to 24-months
Measure: Mean (Standard Error); unit: kg/m^2
Groups:
- Continued Group: Online self-monitoring along with health coach electronic communication and support and real-time updates to primary care physicians
  Health coach electronic communication and support: Health coach reviews responses to weight-related surveys and provides feedback and advice
  Online self-monitoring: Tracking weight, calories, fat grams, and physical activity in electronic personal health record
  Real-time updates to Primary Care physicians: Primary care physicians will receive updates through electronic health record system before each scheduled appointment
Arm/Group | Continued Group | Tracking Group
Number analyzed (Participants) | 80 | 77
kg/m^2 | 0.80 (0.22) | 1.80 (0.23)

3. Secondary Outcome: Waist Circumference (cm)
Description: Waist circumference (cm), change from baseline, Estimate (SE) [95% CI]
Time Frame: Baseline to 24-months
Measure: Mean (Standard Error); unit: centimeters
Arm/Group | Coaching Group | Tracking Group
Number analyzed (Participants) | 80 | 77
centimeters | 1.34 (0.73) | 3.83 (0.74)

4. Secondary Outcome: Maintenance of 5% Weight Loss
Description: Participants maintaining 5% weight loss, No (%)
Time Frame: Baseline to 24-months
Measure: Count of Participants; unit: Participants
Arm/Group | Coaching Group | Tracking Group
Number analyzed (Participants) | 80 | 77
Participants | 79 | 73

5. Secondary Outcome: Pedometer Steps Per Day
Description: Pedometer steps per day, change from baseline, Estimate (SE) [95% CI]
Time Frame: Baseline to 24 months
Measure: Mean (Standard Error); unit: Steps per day
Arm/Group | Coaching Group | Tracking Group
Number analyzed (Participants) | 80 | 77
Steps per day | -335.83 (302.24) | -750.68 (302.76)

6. Secondary Outcome: Physical Component Score (SF-36)
Description: Physical Component score, Estimate (SE) [95% CI] The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Baseline to 24-months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Continued Group | Tracking Group
Number analyzed (Participants) | 80 | 79
score on a scale | -1.95 (0.77) | -3.47 (0.79)

7. Secondary Outcome: Mental Component Score (SF-36)
Description: Mental Component score, Estimate (SE) [95% CI] The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Baseline to 24-months
Measure: Mean (Standard Error); unit: score
Arm/Group | Continued Group | Tracking Group
Number analyzed (Participants) | 80 | 77
score | -2.49 (0.89) | -2.98 (0.09)

8. Secondary Outcome: WOMAC Function Score
Description: WOMAC function score, change from baseline, Estimate (SE) [95% CI] Western Ontario and McMaster Universities Osteoarthritis Index function scale WOMAC function scores are given on a best-to-worst scale of 0-to-100
Time Frame: Baseline to 24 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Continued Group | Tracking Group
Number analyzed (Participants) | 80 | 77
score on a scale | 3.20 (1.17) | 1.22 (1.19)

9. Secondary Outcome: Systolic Blood Pressure
Description: Systolic Blood Pressure (mmHg), change from baseline, Estimate (SE) [95% CI]
Time Frame: Baseline to 24-months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Continued Group | Tracking Group
Number analyzed (Participants) | 80 | 77
mmHg | 4.63 (1.49) | 8.44 (1.53)

10. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic Blood Pressure (mmHg), change from baseline, Estimate (SE) [95% CI]
Time Frame: Baseline to 24-months
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Continued Group | Tracking Group
Number analyzed (Participants) | 80 | 77
mmHg | 2.78 (0.95) | 4.58 (0.98)

11. Other Pre Specified Outcome: Primary Care Provider (PCP) Satisfaction
Description: PCP satisfaction and perceived usefulness of a technologic intervention to improve self-management of patients' weight will be assessed at the end of the first year (12 months) and at the end of the study (30 months).
Time Frame: 12 Months and 30 Months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Patient Satisfaction
Description: Patient satisfaction and perceived usefulness of a technologic intervention to improve self-management of weight will be assessed at the end of the first year (12 months) and the end of the study (30 months).
Time Frame: 12 Months and 30 Months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Dietary Score
Description: Dietary score, change from baseline, Estimate (SE) [95% CI] Dietary score scale is 0-7. Lower scores indicate a diet that is less heart-healthy.
Time Frame: Baseline to 24-months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Continued Group | Tracking Group
Number analyzed (Participants) | 80 | 77
score on a scale | -0.21 (0.14) | -0.23 (0.15)

ADVERSE EVENTS:
Time Frame: 24-months
Description: For adverse medical events, the following guidelines were used to describe severity.
  * Mild
  * Moderate
  * Severe
  Participants were asked about any adverse medical events that might have affected their participation in usual daily activities at each follow-up assessment and self-rated the severity of the event (as opposed to a formal adjudication process).
Arm/Group | Continued Group | Tracking Group
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/96
Other Adverse Events (participants affected / at risk) | 48/98 | 67/96
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continued Group (N=98) | Tracking Group (N=96)
Severe events (General disorders) | 10 (10) | 20 (20) — •Severe - interrupt a participant's usual daily activity. Severe events are usually potentially life-threatening or incapacitating. Of note, the term "severe" does not necessarily equate to "serious"
Moderate (General disorders) | 28 (28) | 33 (33) — Moderate - Events result in a low level of inconvenience or concern with the intervention measures. Moderate events may cause some interference with functioning
Mild (General disorders) | 10 (10) | 14 (14) — •Mild - Events require minimal or no treatment and do not interfere with the participant's daily activities

LIMITATIONS AND CAVEATS:
1)Single-site trial and study population (26%men and 12%non-white) limits generalizability 2)Staff not blinded, leads to some bias in assessment 4)Missing data introduces potential bias in outcomes 5) 24-month endpoint lead to a shorter intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT01946191/Prot_SAP_000.pdf